CLINICAL TRIAL: NCT04525456
Title: Changes in the Immune Responses With Reduxium in Healthy Adults
Brief Title: Immune Responses With Reduxium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ogevity Therapeutics, Inc. (Industry)
Collaborators: National University of Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0101.2006.0101.0001
Record Dates: First submitted 2020-06-29; First posted 2020-08-25 (Actual); Results first posted 2022-05-27 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Immune Tolerance; Viral Infection
Keywords: Antibody; Immunophenotyping; Immune cells
MeSH Terms: conditions — Virus Diseases

STUDY DESIGN:
Intervention Model Description: single-centre, one-arm, prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Reduxium (Experimental): 1 oral drop (0.05ml) per 10kg of body weight (max 8 drops), every 8 hours (3 times a day) for 14 days
  Interventions: Dietary Supplement: Reduxium

INTERVENTIONS:
Dietary Supplement: Reduxium — Single-centre, one-arm, prospective study of 20 healthy subjects who will be given Reduxium supplementation for 14 days.

SUMMARY:
Reduxium is a dietary supplement that provides immune support. This natural compound is orally-ingested in the form of droplets in water to boost the immune system and control inflammation. There is not enough data on the mechanism associated with the action of Reduxium or the extent of the immune response increase it produces. In this study, the investigators propose treating a group of healthy volunteers with Reduxium and investigate the utility of this approach in boosting the native and adaptive immune responses that correlate with immune protection. This may form the basis for a future study employing the product in infectious disease patients.

DETAILED DESCRIPTION:
With the global population increasingly exposed to pandemic crises, permanent and expedient solutions are needed at an affordable cost. Vaccination is less than ideal as the virus is prone to a mutation that renders the previous generation of vaccine less effective. Epidemic and pandemic of viruses infection has become more common and affects both developed and less developed communities. Overcrowding and poor hygiene have been cited to be the major factors in these epidemics, but the host immune system and the ability of the human system to ward off virus infection is a factor less mentioned.

Nutrition is a critical determinant of immune responses and malnutrition the most common cause of immunodeficiency worldwide. Protein-energy malnutrition is associated with a significant impairment of cell-mediated immunity, phagocyte function, complement system, secretory immunoglobulin A antibody concentrations, and cytokine production. Deficiency of single nutrients also results in altered immune responses: this is observed even when the deficiency state is relatively mild. Of the micronutrients, zinc; selenium; iron; copper; vitamins A, C, E, and B6; and folic acid have important influences on immune responses. Adequate intake of vitamins B6, folate, B12, C, E, and of selenium, zinc, copper, and iron supports a T helper cell (Th)1 cytokine-mediated immune response with sufficient production of proinflammatory cytokines, which maintains an effective immune response and avoids a shift to an anti-inflammatory Th2 cell-mediated immune response and an increased risk of extracellular infections. Supplementation with these micronutrients reverses the Th2 cell-mediated immune response to a proinflammatory Th1 cytokine-regulated response with enhanced innate immunity.

Reduxium, a dietary supplement that provides immune support, is a low-cost candidate to boost immune response. Reduxium is a natural compound commercialised in the USA that helps restore homeostasis and controls inflammation. As no toxins or allergens are used, but purely food grade compounds, it is classified as a dietary supplement. Its current purpose is not to treat, diagnose, prevent or cure any disease, but it has immunomodulatory properties. Reduxium is manufactured using a proprietary reactor - a "biochemical cavitation mixer" that allows to create a "smart small molecule". The principal device belongs to the cavitation technology family and is used for the intensification of technological processes in liquid media (liquid processing, splitting of complex molecules, "cold" pasteurization, destruction of solid inclusions). The usage of this process technology enables compression of a set of molecules to 1/12th their original size. Its components are: Phosphoric Acid (58%), Microelement Complex (33.6%) (Zinc, Copper, Iron Pyrophosphate, Potassium, Calcium, Silica, Glycyrrhizic Acid (8.4%). The Microelement Complex is made up of a homogenized complex with special indication, pH =0.0008-0.4, waterless in the final composition.The complex molecules generated scan at the cellular level for the presence of pathogenic (bacterial, viral, fungal) etiologies by reading the characteristics of the electron proton (KNa) pump on the membrane. If these characteristics are violated, the supplement "enters" the cell. At the intra-cellular level, the supplement scans the cell in search of pathology; this "scanning process" is made on the basis of selectivity (healthy - do not touch/ill - induce apoptosis) through the mechanism of mitochondria activity. Specifically, the complex molecules start a cascade of biochemical processes (switching to mitochondria aerobic oxidation, restarting the methyl group with the "epigenetic" effects on DNA, apoptosis). It is unclear how and to which extent this mechanism contributes to innate immune activation following cellular damage and stress, or how it contributes to the adaptive immune response of T and B cells. The primary objective is to analyse the changes in the immune responses after two weeks of Reduxium intake.The secondary objective is to analyse the safety and tolerability of Reduxium.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of 21 - 50 years of age
* Normal blood pressure (BP <140/90 nnHg)
* Normal fasting glucose (<6mmol/L)
* Subjects must stop all supplement for 1 month prior to enrolment

Exclusion Criteria:

* Subjects with known history of lungs or cardiovascular disease
* History of previous pancreatitis
* Past or current history of malignancy
* Subjects with type 2 diabetes
* Past or current history of peptic ulcer disease
* Current pregnancy or breastfeeding

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-01-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Singapore (3):
  - National University of Singapore - The N.1 Institute for Health, Singapore
  - National University of Singapore - Yong Loo Lin School of Medicine, Singapore
  - National University Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available

REFERENCES:
- [Background] Chandra RK. Nutrition and the immune system: an introduction. Am J Clin Nutr. 1997 Aug;66(2):460S-463S. doi: 10.1093/ajcn/66.2.460S. PMID 9250133
- [Background] Wintergerst ES, Maggini S, Hornig DH. Contribution of selected vitamins and trace elements to immune function. Ann Nutr Metab. 2007;51(4):301-23. doi: 10.1159/000107673. Epub 2007 Aug 28. PMID 17726308
- [Background] Cui W, Fan Y, Wu W, Zhang F, Wang JY, Ni AP. Expression of lymphocytes and lymphocyte subsets in patients with severe acute respiratory syndrome. Clin Infect Dis. 2003 Sep 15;37(6):857-9. doi: 10.1086/378587. Epub 2003 Aug 28. PMID 12955652
- [Background] Li T, Qiu Z, Zhang L, Han Y, He W, Liu Z, Ma X, Fan H, Lu W, Xie J, Wang H, Deng G, Wang A. Significant changes of peripheral T lymphocyte subsets in patients with severe acute respiratory syndrome. J Infect Dis. 2004 Feb 15;189(4):648-51. doi: 10.1086/381535. Epub 2004 Feb 4. PMID 14767818

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment happened between October 7, 2020 and January 27, 2021 at National University Hospital (NUH) in Singapore.
Period: Overall Study
Arm/Group | Reduxium
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Reduxium: The intervention consists of 1 oral drop of Reduxium (0.05ml) per 10kg of body weight (max 8 drops), every 8 hours (3 times a day) for 14 days.
Arm/Group | Reduxium
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.4 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Singapore | 20

OUTCOME MEASURES:

1. Primary Outcome: Immune T Cell Subsets and Immunophenotype After 2 Weeks of Reduxium Intake
Description: Blood tests of T cell subsets and phenotypes utilising groups of labelled antibodies
Time Frame: Baseline and weeks 3, 4, 5, 6, 7 and 8 post-baseline
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Reduxium
Number analyzed (Participants) | 20
percentage of cells
  Baseline - Total T cells | 60.53 (9.24)
  Week 3 - Total T cells | 60 (10.27)
  Week 4 - Total T cells | 59.29 (9.44)
  Week 5 - Total T cells | 56.52 (11.88)
  Week 6 - Total T cells | 57.44 (12.75)
  Week 7 - Total T cells | 58.54 (10.23)
  Week 8 - Total T cells | 58.54 (11.09)
  Baseline - Total CD8 (cluster of differentiation 8)+ T cells | 34.08 (8.98)
  Week 3 - Total CD8+ T cells | 35.08 (8.71)
  Week 4 - Total CD8+ T cells | 35.08 (9.19)
  Week 5 - Total CD8+ T cells | 34.46 (9.34)
  Week 6 - Total CD8+ T cells | 35.30 (8.88)
  Week 7 - Total CD8+ T cells | 34.68 (9.93)
  Week 8 - Total CD8+ T cells | 34.49 (9.56)
  Baseline - Exhausted CD8+ T cells | 1.81 (1.15)
  Week 3 - Exhausted CD8+ T cells | 2.06 (1.42)
  Week 4 - Exhausted CD8+ T cells | 2.03 (1.44)
  Week 5 - Exhausted CD8+ T cells | 1.61 (1.00)
  Week 6 - Exhausted CD8+ T cells | 1.78 (1.18)
  Week 7 - Exhausted CD8+ T cells | 2.00 (1.36)
  Week 8 - Exhausted CD8+ T cells | 1.88 (1.08)
  Baseline - Total CD4+ cells | 54.16 (10.98)
  Week 3 - Total CD4+ cells | 53.57 (12.13)
  Week 4 - Total CD4+ cells | 53.97 (11.34)
  Week 5 - Total CD4+ cells | 53.34 (12.22)
  Week 6 - Total CD4+ cells | 53.58 (10.85)
  Week 7 - Total CD4+ cells | 54.79 (12.30)
  Week 8 - Total CD4+ cells | 54.49 (12.54)
  Baseline - Exhausted CD4+ T cells | 11.30 (5.46)
  Week 3 -Exhausted CD4+ T cells | 11.93 (5.39)
  Week 4 -Exhausted CD4+ T cells | 11.15 (4.49)
  Week 5 -Exhausted CD4+ T cells | 10.87 (5.96)
  Week 6 -Exhausted CD4+ T cells | 10.65 (5.15)
  Week 7 -Exhausted CD4+ T cells | 11.59 (5.76)
  Week 8 -Exhausted CD4+ T cells | 11.27 (4.90)
  Baseline -Regulatory T cells (Tregs) | 6.32 (1.39)
  Week 3 - Regulatory T cells (Tregs) | 6.95 (1.50)
  Week 4 - Regulatory T cells (Tregs) | 7.34 (1.80)
  Week 5 - Regulatory T cells (Tregs) | 6.49 (1.93)
  Week 6 - Regulatory T cells (Tregs) | 6.88 (1.90)
  Week 7 - Regulatory T cells (Tregs) | 6.81 (1.90)
  Week 8 - Regulatory T cells (Tregs) | 7.05 (1.53)
  Baseline - chemokine receptor 3 (CXCR3)-Chemokine receptor 6 (CCR6)+ | 1.02 (1.45)
  Week 3 - CXCR3-CCR6+ | 1.24 (2.24)
  Week 4 - CXCR3-CCR6+ | 1.09 (1.81)
  Week 5 - CXCR3-CCR6+ | 1.60 (2.23)
  Week 6 - CXCR3-CCR6+ | 1.34 (1.94)
  Week 7 - CXCR3-CCR6+ | 1.32 (1.92)
  Week 8 - CXCR3-CCR6+ | 1.09 (1.63)
  Baseline - T helper (Th) 1/Th17 cells | 7.17 (5.19)
  Week 3 - Th1/Th17 cells | 6.02 (5.48)
  Week 4 - Th1/Th17 cells | 5.33 (5.12)
  Week 5 - Th1/Th17 cells | 4.55 (3.92)
  Week 6 - Th1/Th17 cells | 4.57 (3.67)
  Week 7 - Th1/Th17 cells | 4.70 (3.69)
  Week 8 - Th1/Th17 cells | 4.56 (3.80)
  Baseline - Th1 cells | 48.63 (24.93)
  Week 3 - Th1 cells | 45.58 (30.23)
  Week 4 - Th1 cells | 44.85 (31.63)
  Week 5 - Th1 cells | 44.15 (31.98)
  Week 6 - Th1 cells | 47.80 (33.09)
  Week 7 - Th1 cells | 47.30 (30.82)
  Week 8 - Th1 cells | 47.58 (32.12)
  Baseline - Th17 cells | 1.28 (0.80)
  Week 3 - Th17 cells | 1.16 (0.91)
  Week 4 - Th17 cells | 1.21 (0.99)
  Week 5 - Th17 cells | 1.19 (1.07)
  Week 6 - Th17 cells | 1.16 (1.16)
  Week 7 - Th17 cells | 1.14 (0.84)
  Week 8 - Th17 cells | 1.24 (1.22)
  Baseline - Th2 cells | 2.86 (1.75)
  Week 3 - Th2 cells | 3.67 (2.28)
  Week 4 - Th2 cells | 3.58 (2.13)
  Week 5 - Th2 cells | 3.46 (1.97)
  Week 6 - Th2 cells | 3.56 (1.94)
  Week 7 - Th2 cells | 3.82 (2.33)
  Week 8 - Th2 cells | 4.05 (2.23)
  Baseline - T follicular helper cells (Tfh) | 13.75 (2.67)
  Week 3 - T follicular helper cells (Tfh) | 12.75 (3.52)
  Week 4 - T follicular helper cells (Tfh) | 12.02 (3.48)
  Week 5 - T follicular helper cells (Tfh) | 12.40 (3.83)
  Week 6 - T follicular helper cells (Tfh) | 12.22 (3.16)
  Week 7 - T follicular helper cells (Tfh) | 12.33 (3.50)
  Week 8 - T follicular helper cells (Tfh) | 11.58 (4.92)
  Baseline - Activated Tfh (Inducible T-cell Costimulator (ICOS+)) | 0.50 (0.24)
  Week 3 - Activated Tfh (ICOS+) | 0.45 (0.24)
  Week 4 - Activated Tfh (ICOS+) | 0.44 (0.27)
  Week 5 - Activated Tfh (ICOS+) | 0.38 (0.22)
  Week 6 - Activated Tfh (ICOS+) | 0.40 (0.23)
  Week 7 - Activated Tfh (ICOS+) | 0.47 (0.26)
  Week 8 - Activated Tfh (ICOS+) | 0.48 (0.32)
  Baseline - Activated Tfh (Programmed cell death protein 1 (PD-1+)) | 2.30 (0.84)
  Week 3 - Activated Tfh (PD-1+) | 2.25 (0.88)
  Week 4 - Activated Tfh (PD-1+) | 2.08 (1.01)
  Week 5 - Activated Tfh (PD-1+) | 2.01 (0.85)
  Week 6 - Activated Tfh (PD-1+) | 2.08 (0.85)
  Week 7 - Activated Tfh (PD-1+) | 2.20 (0.91)
  Week 8 - Activated Tfh (PD-1+) | 2.18 (1.16)
  Baseline - Activated Tfh (ICOS+PD-1+) | 1.18 (0.67)
  Week 3 - Activated Tfh (ICOS+PD-1+) | 1.17 (0.58)
  Week 4 - Activated Tfh (ICOS+PD-1+) | 1.18 (0.60)
  Week 5 - Activated Tfh (ICOS+PD-1+) | 1.00 (0.49)
  Week 6 - Activated Tfh (ICOS+PD-1+) | 1.08 (0.46)
  Week 7 - Activated Tfh (ICOS+PD-1+) | 1.32 (0.89)
  Week 8 - Activated Tfh (ICOS+PD-1+) | 1.33 (0.84)

2. Primary Outcome: Immune B Cell Subsets and Immunophenotype After 2 Weeks of Reduxium Intake
Description: Blood tests of B cell subsets and phenotypes utilising groups of labelled antibodies
Time Frame: Baseline and weeks 3, 4, 5, 6, 7 and 8 post-baseline
Population: healthy participants
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Reduxium
Number analyzed (Participants) | 20
percentage of cells
  Baseline - Total B cells | 17.44 (6.89)
  Week 3 - Total B cells | 21.09 (12.68)
  Week 4 - Total B cells | 18.64 (7.32)
  Week 5 - Total B cells | 19.84 (10.33)
  Week 6 - Total B cells | 20.70 (9.28)
  Week 7 - Total B cells | 20.48 (8.92)
  Week 8 - Total B cells | 22.05 (10.99)
  Baseline - Memory B cells (MBCs) | 7.47 (3.18)
  Week 3 - Memory B cells (MBCs) | 7.34 (3.08)
  Week 4 - Memory B cells (MBCs) | 7.63 (3.91)
  Week 5 - Memory B cells (MBCs) | 7.44 (3.46)
  Week 6 - Memory B cells (MBCs) | 7.17 (2.93)
  Week 7 - Memory B cells (MBCs) | 7.53 (3.38)
  Week 8 - Memory B cells (MBCs) | 7.66 (3.68)
  Baseline - Classical MBCs | 1.24 (0.78)
  Week 3 - Classical MBCs | 0.96 (0.55)
  Week 4 - Classical MBCs | 1.06 (0.69)
  Week 5 - Classical MBCs | 1.15 (0.60)
  Week 6 - Classical MBCs | 0.90 (0.48)
  Week 7 - Classical MBCs | 0.91 (0.53)
  Week 8 - Classical MBCs | 0.93 (0.57)
  Baseline - Activated MBCs | 6.28 (2.78)
  Week 3 - Activated MBCs | 6.37 (2.79)
  Week 4 - Activated MBCs | 6.59 (3.69)
  Week 5 - Activated MBCs | 6.46 (3.15)
  Week 6 - Activated MBCs | 6.25 (2.69)
  Week 7 - Activated MBCs | 6.61 (3.09)
  Week 8 - Activated MBCs | 6.71 (3.38)
  Baseline - Tissue-like MBCs | 1.27 (0.90)
  Week 3 - Tissue-like MBCs | 1.01 (0.62)
  Week 4 - Tissue-like MBCs | 1.09 (0.69)
  Week 5 - Tissue-like MBCs | 1.04 (0.63)
  Week 6 - Tissue-like MBCs | 0.96 (0.56)
  Week 7 - Tissue-like MBCs | 0.95 (0.54)
  Week 8 - Tissue-like MBCs | 0.99 (0.60)
  Baseline - Switched B cells | 1.58 (1.24)
  Week 3 - Switched B cells | 1.23 (1.21)
  Week 4 - Switched B cells | 1.39 (1.21)
  Week 5 - Switched B cells | 1.33 (1.12)
  Week 6 - Switched B cells | 1.17 (1.06)
  Week 7 - Switched B cells | 1.35 (1.13)
  Week 8 - Switched B cells | 1.75 (2.15)
  Baseline - Unswitched B cells | 7.96 (3.37)
  Week 3 - Unswitched B cells | 7.76 (3.26)
  Week 4 - Unswitched B cells | 8.16 (4.27)
  Week 5 - Unswitched B cells | 7.90 (3.60)
  Week 6 - Unswitched B cells | 7.58 (3.07)
  Week 7 - Unswitched B cells | 7.98 (3.52)
  Week 8 - Unswitched B cells | 8.11 (3.83)
  Baseline - Naïve B cells | 4.74 (2.61)
  Week 3 - Naïve B cells | 5.13 (3.00)
  Week 4 - Naïve B cells | 5.02 (3.02)
  Week 5 - Naïve B cells | 4.85 (3.07)
  Week 6 - Naïve B cells | 4.97 (3.10)
  Week 7 - Naïve B cells | 5.28 (3.18)
  Week 8 - Naïve B cells | 5.55 (3.41)
  Baseline - Plasmablasts | 5.38 (3.63)
  Week 3 - Plasmablasts | 4.67 (3.79)
  Week 4 - Plasmablasts | 4.85 (3.68)
  Week 5 - Plasmablasts | 5.12 (3.89)
  Week 6 - Plasmablasts | 4.66 (3.53)
  Week 7 - Plasmablasts | 4.21 (3.08)
  Week 8 - Plasmablasts | 4.33 (3.26)
  Baseline - Exhausted B cells | 3.13 (1.83)
  Week 3 - Exhausted B cells | 2.36 (1.48)
  Week 4 - Exhausted B cells | 2.68 (1.88)
  Week 5 - Exhausted B cells | 2.71 (1.50)
  Week 6 - Exhausted B cells | 2.25 (1.22)
  Week 7 - Exhausted B cells | 2.45 (1.33)
  Week 8 - Exhausted B cells | 2.83 (2.31)

3. Primary Outcome: Innate Immune Cell Subsets (Monocytes -Cluster of Differentiation 14 R-Phycoerythrin (CD14PE)) After 2 Weeks of Reduxium Intake
Description: Blood tests of monocytes subsets utilising groups of labelled antibodies
Time Frame: Baseline and weeks 3, 4, 5, 6, 7 and 8 post-baseline
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Reduxium
Number analyzed (Participants) | 20
percentage of cells
  Baseline - Non-classical monocytes | 4.88 (3.41)
  Week 3 - Non-classical monocytes | 2.50 (1.84)
  Week 4 - Non-classical monocytes | 2.99 (2.01)
  Week 5 - Non-classical monocytes | 2.94 (2.15)
  Week 6 - Non-classical monocytes | 2.51 (2.04)
  Week 7 - Non-classical monocytes | 2.73 (1.80)
  Week 8 - Non-classical monocytes | 3.26 (1.68)
  Baseline - Intermediate monocytes | 7.26 (7.17)
  Week 3 - Intermediate monocytes | 4.00 (5.63)
  Week 4 - Intermediate monocytes | 5.60 (5.60)
  Week 5 - Intermediate monocytes | 5.79 (7.20)
  Week 6 - Intermediate monocytes | 5.41 (6.23)
  Week 7 - Intermediate monocytes | 6.08 (6.32)
  Week 8 - Intermediate monocytes | 7.49 (7.31)
  Baseline - Classical monocytes | 78.92 (11.78)
  Week 3 - Classical monocytes | 84.86 (8.92)
  Week 4 - Classical monocytes | 83.27 (9.06)
  Week 5 - Classical monocytes | 83.68 (10.25)
  Week 6 - Classical monocytes | 85.39 (8.31)
  Week 7 - Classical monocytes | 84.87 (8.45)
  Week 8 - Classical monocytes | 82.72 (10.86)

4. Primary Outcome: Innate Immune Cell Subsets [Natural Killer (NK) Cells (CD56 Allophycocyanin (APC)] After 2 Weeks of Reduxium Intake
Description: Blood tests of NK cell subsets utilising groups of labelled antibodies
Time Frame: Baseline and weeks 3, 4, 5, 6, 7 and 8 post-baseline
Population: healthy participants.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Reduxium
Number analyzed (Participants) | 20
percentage of cells
  CD16++CD56- - Baseline | 0.89 (0.62)
  Week 3 - CD16++CD56- | 0.91 (0.50)
  Week 4 - CD16++CD56- | 0.99 (0.44)
  Week 5 - CD16++CD56- | 0.83 (0.39)
  Week 6 - CD16++CD56- | 1.02 (0.58)
  Week 7 - CD16++CD56- | 1.24 (0.60)
  Week 8 - CD16++CD56- | 1.34 (0.56)
  Baseline - CD16+CD56+ | 67.89 (13.20)
  Week 3 - CD16+CD56+ | 66.63 (15.26)
  Week 4 - CD16+CD56+ | 66.31 (15.48)
  Week 5 - CD16+CD56+ | 67.07 (15.67)
  Week 6 - CD16+CD56+ | 69.92 (13.13)
  Week 7 - CD16+CD56+ | 69.86 (10.90)
  Week 8 - CD16+CD56+ | 69.04 (13.01)
  Baseline - CD16+CD56++ | 0.94 (0.47)
  Week 3 - CD16+CD56++ | 1.09 (0.68)
  Week 4 - CD16+CD56++ | 0.96 (0.45)
  Week 5 - CD16+CD56++ | 0.90 (0.42)
  Week 6 - CD16+CD56++ | 1.08 (0.59)
  Week 7 - CD16+CD56++ | 1.06 (0.45)
  Week 8 - CD16+CD56++ | 1.23 (0.68)
  Baseline - CD16-CD56+ | 2.05 (1.01)
  Week 3 - CD16-CD56+ | 1.78 (0.98)
  Week 4 - CD16-CD56+ | 1.68 (0.69)
  Week 5 - CD16-CD56+ | 1.68 (0.84)
  Week 6 - CD16-CD56+ | 1.61 (0.73)
  Week 7 - CD16-CD56+ | 1.66 (0.73)
  Week 8 - CD16-CD56+ | 1.56 (0.84)
  Baseline - CD16-CD56++ | 2.98 (1.54)
  Week 3 - CD16-CD56++ | 2.90 (1.60)
  Week 4 - CD16-CD56++ | 2.66 (1.23)
  Week 5 - CD16-CD56++ | 2.61 (1.26)
  Week 6 - CD16-CD56++ | 2.84 (1.44)
  Week 7 - CD16-CD56++ | 2.67 (1.06)
  Week 8 - CD16-CD56++ | 3.16 (1.79)

5. Primary Outcome: Renal Panel (Sodium) After 2 Weeks of Reduxium Intake
Description: Sodium blood tests
Time Frame: Baseline and week 8 post-baseline
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Reduxium
Number analyzed (Participants) | 20
mmol/L
  Baseline | 139.55 (1.43)
  Week 8 | 139.40 (1.59)

6. Primary Outcome: Renal Panel (Potassium) After 2 Weeks of Reduxium Intake
Description: Potassium blood tests
Time Frame: Baseline and week 8 post-baseline
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Reduxium
Number analyzed (Participants) | 20
mmol/L
  Baseline | 4.26 (0.49)
  Week 8 | 4.54 (0.46)

7. Primary Outcome: Renal Panel (Urea) After 2 Weeks of Reduxium Intake
Description: Urea blood tests
Time Frame: Baseline and week 8 post-baseline
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Reduxium
Number analyzed (Participants) | 20
mmol/L
  Baseline | 4.20 (1.45)
  Week 8 | 4.04 (1.08)

8. Primary Outcome: Renal Panel (Creatinine) After 2 Weeks of Reduxium Intake
Description: Creatinine blood tests
Time Frame: Baseline and week 8 post-baseline
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Reduxium
Number analyzed (Participants) | 20
umol/L
  Baseline | 69.05 (12.09)
  Week 8 | 68.85 (11.76)

9. Primary Outcome: Liver Panel (Aspartate Aminotransferase (AST)) After 2 Weeks of Reduxium Intake
Description: AST blood tests
Time Frame: Baseline and week 8 post-baseline
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Reduxium
Number analyzed (Participants) | 20
U/L
  Baseline | 19.50 (3.35)
  Week 8 | 20.55 (4.15)

10. Primary Outcome: Liver Panel (Alanine Aminotransferase (ALT)) After 2 Weeks of Reduxium Intake
Description: ALT blood tests
Time Frame: Baseline and week 8 post-baseline
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Reduxium
Number analyzed (Participants) | 20
U/L
  Baseline | 15.90 (7.66)
  Week 8 | 17.40 (9.45)

11. Primary Outcome: Liver Panel (Albumin) After 2 Weeks of Reduxium Intake
Description: Albumin blood tests
Time Frame: Baseline and week 8 post-baseline
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Reduxium
Number analyzed (Participants) | 20
g/L
  Baseline | 42.80 (3.37)
  Week 8 | 42.95 (2.03)

12. Primary Outcome: Liver Panel (Alkaline Phosphatase (ALP)) After 2 Weeks of Reduxium Intake
Description: ALP blood tests
Time Frame: Baseline and week 8 post-baseline
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Reduxium
Number analyzed (Participants) | 20
U/L
  Baseline | 62.90 (19.82)
  Week 8 | 59.90 (15.87)

13. Primary Outcome: Liver Panel (Bilirubin) After 2 Weeks of Reduxium Intake
Description: Bilirubin blood tests
Time Frame: Baseline and week 8 post-baseline
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Reduxium
Number analyzed (Participants) | 20
umol/L
  Baseline | 11.90 (4.09)
  Week 8 | 11.25 (3.50)

14. Primary Outcome: Liver Panel (Lactate Dehydrogenase (LDH)) After 2 Weeks of Reduxium Intake
Description: LDH blood tests
Time Frame: Baseline and week 8 post-baseline
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Reduxium
Number analyzed (Participants) | 20
U/L
  Baseline | 310.80 (43.87)
  Week 8 | 377 (108.54)

15. Secondary Outcome: Number of Adverse Events After Reduxium Intake
Description: To analyse the safety and tolerability of Reduxium after 2 weeks of Reduxium intake, based on number of adverse events
Time Frame: Baseline and weeks 3, 4, 5, 6, 7 and 8 post-baseline
Measure: Number; unit: adverse events
Arm/Group | Reduxium
Number analyzed (Participants) | 20
adverse events | 0

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Reduxium
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol (2020-05-11): https://cdn.clinicaltrials.gov/large-docs/56/NCT04525456/Prot_000.pdf